CLINICAL TRIAL: NCT01131715
Title: Pharmacist Follow-up of Patients With Coronary Heart Disease. A Qualitative Study of Patient Experience.
Brief Title: Pharmacist Follow-up, a Qualitative Study of Patient Experience
Status: Completed | Type: Observational
Sponsor: Hospital Pharmacy of North Norway Trust (Other)
Collaborators: University of Tromso (Other)
Responsible Party: Principal Investigator, Beate Hennie Garcia, PhD, Associate Professor, Hospital Pharmacy of North Norway Trust
Other Study IDs: SHAN-002
Record Dates: First submitted 2010-04-30; First posted 2010-05-27 (Estimated); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Patient Satisfaction; Patient Preference
Keywords: Qualitetive interview; Coronary heart disease (CHD); Patient experience; Patient perception
MeSH Terms: conditions — Patient Satisfaction; Patient Preference; Coronary Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study group: Patients who are included in the pharmacist follow-up procedure

SUMMARY:
A pharmacist follow-up procedure is under development. Patients with coronary heart disease (CHD) is being followed up by a pharmacist for one year with three meetings; at discharge from hospital, after three months and after one year. The evaluation is basically based on quantitative measures as achievement of therapeutic goals, number of drug related problems detected, hospitalisations etc. However, the patients' own experience with the follow-up procedure cannot be evaluated using these measures. Thus, a qualitative approach is needed. In this study, a total of four patients participating in the follow-up will be included and interviewed. A semistructured interview guide will be used. Interviews will be taped, transcribed and analyzed with the intention to explore how patients experience the follow-up from the pharmacist. A thoruough content analysis will be performed. Patients included must have met the pharmacist at least twice. The pharmacist in charge of the follow-up will recruit patients and hand out study information. Patients will reply to the principal investigator of the study and thus kept anonymous for the pharmacist in charge of the follow-up. No pressure will be put on the patients to join, but it will be emphasized that it will help evaluating the procedure.

DETAILED DESCRIPTION:
See full publication on http://www.biomedcentral.com/1756-0500/7/197 Garcia et al. BMC Research Notes 2014, 7:197

ELIGIBILITY:
Inclusion Criteria:

* must have met the pharmacist at least twice
* living within the area of Tromsoe city so that interviews are possible

Exclusion Criteria

* none as patients are already enrolled in another study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in the study "Pharmacist follow-up of patients with CHD".
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2010-03 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Qualitative evaluation of the impact of pharmacist follow-up via interviews with the participating patients | 3 months or 1 year
  In the pharmacist follow-up procedure under development, patients have individual "consultations" with a pharmacist three times. Patients are recruited to this study at the second or third consultation. Interviews will be performed with patients included to explore how patients' experience this follow-up procedure. Outcome measures from patient interviews can be counted. In qualitative research, the content of the interviews are thoroughly analysed with focus on the meaning of the informant's/interviewee's sayings. Outcomes will be presented as overall themes touched by the informants.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Smaabrekke, PhD, Principal Investigator — University of Tromso; Beate H Garcia, PhD, Study Chair — Hospital Pharmacy of North Norway Trust
Locations (1):
- University of Tromsoe, Tromsø, Norway

REFERENCES:
- [Derived] Garcia BH, Storli SL, Smabrekke L. A pharmacist-led follow-up program for patients with coronary heart disease in North Norway--a qualitative study exploring patient experiences. BMC Res Notes. 2014 Mar 29;7:197. doi: 10.1186/1756-0500-7-197. PMID 24679131
- See also: Published article — http://www.biomedcentral.com/1756-0500/7/197